CLINICAL TRIAL: NCT04925427
Title: Justice Community Opioid Innovation Network (JCOIN): Reducing Opioid Mortality in Illinois
Brief Title: Reducing Opioid Mortality in Illinois
Acronym: ROMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Community Outreach Intervention Projects (Unknown); Cook County Sheriff Office (Unknown); Cook County Health & Hospitals System (Other); Lake County Sheriff Office (Unknown); LaSalle County Jail (Unknown); Perfectly Flawed Foundation (Unknown); Jackson County Sheriff Office (Unknown); Illinois Department of Corrections (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB19-1775
Record Dates: First submitted 2021-05-05; First posted 2021-06-14 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Management and Peer Recovery (Experimental): Participants in the CM/PRC + OEND arm will receive one year of service delivery. During the initial intake interview the CM will identify primary, secondary, and tertiary barriers to treatment initiation and completion, then create an action plan tailored to each client. PRCs with lived SUD or incarceration experience will address recovery barriers, while CMs will focus on service barriers. Where beneficial and desired by the clients, PRCs will accompany clients to provider and select service appointments to promote engagement and retention. CM/PRC teams will provide OEND upon community re-entry. The teams will provide follow-up phone calls and home visits to facilitate service linkages. Contact frequency will depend on clients' individual barriers (e.g., transportation, homelessness), but will include at least weekly in-person or telephone check-ins for first six months, reduced to monthly check-ins after that.
  Interventions: Behavioral: Case Management and Peer Recovery
- Naloxone-Only (Placebo Comparator): Participants randomized to the Usual care + OEND condition will be trained on naloxone administration by research staff at the time of randomization. Upon community re-entry,they will be given a naloxone kit and information on local resources for harm reduction, SUD treatment, and additional supportive services.
  Interventions: Behavioral: Naloxone-Only

INTERVENTIONS:
Behavioral: Case Management and Peer Recovery — A blend between a Critical Time Intervention (CTI) case management model and a peer recovery coaching approach. CORI will employ peer-based case management/recovery coaching and other transitional services (e.g., peer navigation) to provide support and service linkages to medication-assisted treatment (MAT) and harm reduction interventions to reduce subsequent opioid use and related harms.
  Arms: Case Management and Peer Recovery
Behavioral: Naloxone-Only — Participants will be trained on naloxone administration, and upon re-entry, they will be given a naloxone kit and information on local resources for harm reduction, SUD treatment, and additional supportive services.
  Arms: Naloxone-Only

SUMMARY:
Reducing Opioid Mortality in Illinois (ROMI) is 5-year research study led by the University of Chicago in partnership with the University of Illinois at Chicago's (UIC) Community Outreach Intervention Projects (COIP), the Illinois Criminal Justice Information Authority (ICJIA) and the American Institutes for Research (AIR). ROMI aims to understand and test strategies for linking individuals with a history of opioid use disorder who are released from Illinois jails and prisons to substance use treatment. ROMI is one of twelve grants awarded by the National Institutes of Health (NIH) as part of the Justice Community Opioid Innovation Network (JCOIN) to support research on quality addiction treatment for opioid use disorder in criminal justice settings nationwide.

DETAILED DESCRIPTION:
This NIDA-funded multi-site randomized control trial (RCT) examines the effectiveness of an established, intensive case management model for study participants who are awaiting release from four jails and two prisons across Illinois. The investigators seek to demonstrate that a unified case management approach can improve treatment engagement and retention among individuals who face high risks of opioid use disorders, overdose, and related harms. The investigators will examine the impact of case management and peer recovery coaching on participants' engagement with treatment and harm reduction interventions. The investigators will also study secondary outcomes including insurance enrollment, re-arrest, use of mental health services, and more.

ROMI will enroll at least 300 individuals with opioid disorders in the CMPR group, and at least 300 participants in the naloxone-only across five geographically distinct sites of care. All participants will receive harm reduction resources. The investigators hypothesize that the treatment group will display declines in opioid use, re-arrest, self-reported syringe sharing, and overdose risk behaviors relative to the control groups. The investigators will also examine differences between urban - rural and rural differences in treatment engagement and retention engagement, retention, and downstream outcomes across treatment arms. Aside from demonstrating these treatment impacts, the investigators will guide, document and evaluate ROMI's implementation efforts to ensure consistency across sites across sites and to inform future replication of the model in different settings or for different populations. (Edited 11/27/23 to reflect changes in recruitment from 500 in each treatment arm to 300)

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old
* Reside in designated research site county or zip code
* Satisfy criteria for likely OUD based upon nonmedical use of prescription opioids, heroin, or synthetic opioids.

Exclusion Criteria:

* Participants experiencing cognitive impairments that preclude informed consent.
* Reside out of the service area.
* Prior enrollment in a parallel JCOIN study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Addiction treatment engagement | 12 months
  Number (%) of participants with two or more addiction treatment provider encounters within three months of study enrollment

SECONDARY OUTCOMES:
Percent of participants enrolled in Medicaid or private insurance | 12 months
  Defined as Medicaid or private insurance enrollment during the intervention period.
Percent of participant utilizing mental health services | 90 days
  Defined as any mental health utilization within 90 days conditional on CAT-MH diagnostic.
Days of Opioid Use | 12 months
  A self-reported count 0 to 90 days of using any kind of opioids each quarter, as indicated by the Global Appraisal of Individual Needs (GAIN)assessment tool.
Days of stimulant Use | 12 months
  A self-reported count 0 to 90 days of using any kind of stimulants each quarter, as indicated by the Global Appraisal of Individual Needs (GAIN)assessment tool.
Opioid Use Disorder (OUD) Symptoms | 12 months
  A self-reported count of Opioid Use Disorder (OUD) symptoms, again as captured by the GAIN instrument, measuring past month, past 90 days, year, and lifetime. SUD/MH symptoms as captured by the CAT-MH/SUD.
Stimulant Use Disorder Symptoms | 12 months
  A self-reported count of Stimulant Use Disorder symptoms, again as captured by the GAIN instrument, measuring past month, past 90 days, year, and lifetime. SUD/MH symptoms as captured by the CAT-MH/SUD.
Patient Reported Outcomes Measurement Information System | 12 months
  This scale of person-centered measures includes eight domains (physical function, ability to participate in social roles and activities, anxiety, depression, fatigue, sleep disturbance, cognitive function ability, pain interference, and pain intensity). These are elicited in a five point likert scale (from 1= never to 5 = always) with higher scores equaling more of the concept being measured, which may be better or worse based on the domain measured.
Health services costs | 12 months
  This cost measure is based on the self-reported frequency of all healthcare services use. Measured using published Medicare reimbursement rates for all pertinent medical care services. Addiction services cost as measured by DATCAP methodology.
Re-arrest and Re-incarceration | 12 months
  Arrest or re-incarceration based on any charge using data from Illinois Criminal Justice Information Authority (ICJIA). The investigators will examine the binary outcomes of re-arrest and reincarceration, and also count data models of the number of arrests post-enrollment during days of non-incarceration.
Self-reported rate of illegal activity | 12 months
  This is a self-reported count of 19 items across different types of illegal activities following the JCOIN core measures instrument.
Social cost of self reported crime | 12 months
  Total social cost of self-reported illegal activity, using estimates for offense-specific economic valuations of social cost per offense and a self-reported count of 19 items across different types of illegal activities.
Social cost of re-arrest and associated offenses | 12 months
  Total social cost of crime, using estimates for offense-specific economic valuations of social cost per offense and any charge using data from Illinois Criminal Justice Information Authority (ICJIA).
All-cause mortality | 12 months
  Mortality from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Harold Pollack, PhD, Principal Investigator — University of Chicago; Mai Pho, MD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - Cook County Department of Corrections, Chicago, Illinois
  - Jackson County Jail, Murphysboro, Illinois
  - LaSalle County Jail, Ottawa, Illinois
  - Illinois Department of Corrections, Springfield, Illinois
  - Lake County Sheriff's Office Corrections Division, Waukegan, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Will adhere to NIH JCOIN approved plan
Supporting Information: Study Protocol, ICF
Time Frame: Will adhere to NIH JCOIN approved plan
Access Criteria: Will adhere to NIH JCOIN approved plan

REFERENCES:
- [Derived] Pho MT, Bouris A, Carreon ED, Stinnette M, Kaufmann M, Shuman V, Watson DP, Jimenez AD, Powell B, Kaplan C, Zawacki S, Morris S, Garcia J, Hafertepe A, Hafertepe K, Pollack HA, Schneider JA, Boodram B. Implementation strategies to support recovery support workers serving criminal legal involved people who use drugs. J Subst Use Addict Treat. 2025 Feb;169:209583. doi: 10.1016/j.josat.2024.209583. Epub 2024 Nov 23. PMID 39586354